CLINICAL TRIAL: NCT04273763
Title: Evaluating the Efficacy and Safety of Bromhexine Hydrochloride Tablets Combined With Standard Treatment/ Standard Treatment in Patients With Suspected and Mild Novel Coronavirus Pneumonia (COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019NCP1.0
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Novel Coronavirus Pneumonia; 2019-nCoV
MeSH Terms: interventions — Bromhexine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Treatment group
  Interventions: Drug: Bromhexine Hydrochloride Tablets; Drug: Arbidol Hydrochloride Granules; Drug: Recombinant Human Interferon α2b Spray
- Group B (Active Comparator): Control group
  Interventions: Drug: Arbidol Hydrochloride Granules; Drug: Recombinant Human Interferon α2b Spray

INTERVENTIONS:
Drug: Bromhexine Hydrochloride Tablets — Bromhexine Hydrochloride Tablets
  Arms: Group A
Drug: Arbidol Hydrochloride Granules — Standard treatment refers to the latest edition of Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection. Arbidol Hydrochloride Granules is recommended but not enforced to use.
Drug: Recombinant Human Interferon α2b Spray — Standard treatment refers to the latest edition of Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection.

SUMMARY:
Compare the efficacy and safety of Bromhexine Hydrochloride Tablets combined with standard treatment/ standard treatment in patients with suspected and mild, or common novel coronavirus pneumonia (COVID-19).

Random, open, group sequential design.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years (Including 18and 80years, male or female).
* One of them:

  1. Laboratory (RT-PCR) and clinical symptoms confirmed case of novel coronavirus pneumonia (COVID-19).
  2. Patients diagnosed clinically as suspected cases.
* Ability to communicate well with researchers and sign the informed consent Form (ICF) voluntarily.

Exclusion Criteria:

* ALT≥5 times of ULN, level of total bilirubin≥3 times of ULN, or Cr≥1.5 times of ULN.
* Patients with serious severe liver disease.
* Excluded who diagnosed as pneumonia patients with novel coronavirus infection of severe type and critical type. 【Diagnostic criteria reference the official guideline "Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 5) "】.
* Patients with previous history of severe gastrointestinal diseases such as gastric ulcers and bleeding.
* Patients with lactose intolerance.
* Patients who are allergic to the components of this medicine (Major components: Bromhexine Hydrochloride; excipient: starch, lactose, magnesium stearate).
* Positive serum pregnancy test result for women with childbearing potential at screening or lactating women.
* Other circumstances that the researcher considers inappropriate to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2020-05-10 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery after treatment | within 14 days from the start of medication
  Defined as random to fever, respiratory rate return to normal and cough remission over 48 hours.
Rate of aggravation | within 14 days from the start of medication
  Aggravation was defined as(one of them): respiratory distress, RR ≥ 30 times / min; SpO2 ≤ 93% in resting state; arterial partial pressure of oxygen (PaO2) /concentration of oxygen (FiO2) ≤ 300mmHg

SECONDARY OUTCOMES:
Clinical remission rate | within 14 days from the start of medication
  Clinical remission was defined as (one of them): sustained (more than 48 hours) alleviation of illness based on symptom (fever, cough, dyspnea, myalgia, diarrhea and so on) all being absent and no evidence for progression.
Dynamic changes of oxygenation index | within 14 days from the start of medication
  oxygenation index
Time to cure | within 14 days from the start of medication
  time of Clinical recovery, negative COVID-19 nucleic acid results and CT recovery
rate to cure | within 14 days from the start of medication
  proportion of Clinical recovery, negative COVID-19 nucleic acid results and CT recovery among infected patients
Time to defervescence | within 14 days from the start of medication
  defervescence is defined as below 37 Celcius degrees（ear temperature）
Time to cough remission | within 14 days from the start of medication
Time to dyspnea remission | within 14 days from the start of medication
Days of supplemental oxygenation | within 14 days from the start of medication
Rate of patients with requring supplemental oxygen | within 14 days from the start of medication
Rate of patients with mechanical ventilation | within 14 days from the start of medication
Time of negative COVID-19 nucleic acid results | within 14 days from the start of medication
Rate of negative COVID-19 nucleic acid results | within 14 days from the start of medication
Rate of ICU admission | within 14 days from the start of medication
28-day mortality | From the first day of screening to the day of follow-up (28 days)

CONTACTS AND LOCATIONS:
Overall Officials: XIAN SHEN, phd, Study Chair — The 2nd Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second AffIliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No